CLINICAL TRIAL: NCT07172061
Title: Sigh in Pressure Support Ventilation to Detect Respiratory System Compliance and Lung Recruitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Collaborators: Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Principal Investigator, Luca Bastia, MD, AUSL Romagna Rimini
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SIREC
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation
Keywords: Assisted ventilation; Pressure support ventilation (PSV); PEEP; Recruitment; Sigh; Respiratory system compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical PEEP (baseline) (Experimental): Pressure support ventilation (PSV) at the clinical PEEP with ventilator-delivered sighs: one sustained inflation at 30 cmH₂O for 3 seconds every minute.
  Interventions: Other: PSV + sigh (Clinical PEEP and Clinical PEEP + 3 cmH₂O)
- Clinical PEEP +3 cmH₂O (Experimental): Pressure support ventilation (PSV) with PEEP set 3 cmH₂O above the clinical PEEP, with ventilator-delivered sighs: one sustained inflation at 30 cmH₂O for 3 seconds every minute.
  Interventions: Other: PSV + sigh (Clinical PEEP and Clinical PEEP + 3 cmH₂O)

INTERVENTIONS:
Other: PSV + sigh (Clinical PEEP and Clinical PEEP + 3 cmH₂O) — Each patient undergoes two sequential 15-minute steps: 1) pressure support ventilation at the clinical PEEP and 2) the same settings with PEEP increased by 3 cmH₂O. A ventilator-delivered sigh is programmed as one sustained inflation at 30 cmH₂O for 3 seconds every minute. All other ventilator parameters (trigger sensitivity, pressure support level, mandatory breath timing) remain unchanged. At the end of each step, inspiratory and expiratory holds are performed to collect respiratory mechanics and arterial blood gases; compliance during the sigh is calculated once flow is zero and airway pressure is stable.

SUMMARY:
The goal of this physiological study is to determine whether ventilator-delivered sigh breaths during pressure support ventilation (PSV) provide a reliable bedside index of lung recruitability and can guide PEEP optimization.The main questions it aims to answer are:

* Does respiratory system compliance measured at the end of a sigh (Crs_sigh) differ from compliance obtained with an inspiratory hold during an assisted breath (Crs_assisted), and can the Crs_sigh/Crs_assisted ratio indicate recruitability?
* Does adjusting PEEP based on the sigh-derived recruitability index improve respiratory mechanics and gas exchange compared with usual clinical PEEP settings?

DETAILED DESCRIPTION:
Background and RationaleInvasive mechanical ventilation is often necessary in critically ill adults but may contribute to ventilator-induced lung injury (VILI) if ventilator settings are not individualized. During assisted ventilation (pressure support ventilation, PSV), ongoing patient effort complicates the assessment of PEEP response, PEEP titration, and lung recruitability.Ventilator-delivered sigh breaths (i.e., brief sustained inflations) can improve gas exchange and promote alveolar recruitment, and may permit artifact-free assessment of respiratory mechanics in assisted modes. This study evaluates whether Crs measured at the end of a sigh provides reliable, clinically useful information on recruitability and whether the ratio of Crs during sigh to Crs during an assisted breath (Crs_sigh/Crs_assisted) can guide positive end-expiratory pressure (PEEP) optimization.Primary ObjectiveTo assess lung recruitability during PSV by normalizing Crs measured at the end of a sigh to Crs obtained with an inspiratory hold during an assisted breath.Secondary Objectives

* To quantify the proportion of patients in whom Pplat during assisted breathing is not reliable (non-readable or unstable ≥3 s).
* To determine whether adjusting PEEP according to the sigh-derived recruitability index improves Crs.

Inclusion criteria:Adults (≥18 years) receiving PSV with the ventilator's sigh function active.Exclusion criteria:

* Clinical contraindication to increasing PEEP
* Hemodynamic instability defined as SOFA cardiovascular score ≥3

Protocol OverviewEach participant undergoes two sequential, non-randomized steps:

* Step 1 (Clinical PEEP): Measurements are performed after ≥15 minutes at the treating team's current PEEP.
* Step 2 (Clinical PEEP +3 cmH₂O): PEEP is increased by 3 cmH₂O; measurements are repeated after ≥15 minutes of stabilization.

In both steps, a sigh is programmed as a sustained inflation at 30 cmH₂O for 3 seconds (pressure-controlled), per routine practice and prior literature.Sigh Setting

* Sigh frequency: 1 sustained inflation every minute.
* Sigh target: 30 cmH₂O for 3 seconds.
* If end-inspiratory flow did not reach 0 L/min, the inspiratory time of the sigh was extended to ensure an end-inspiratory alveolar pressure of 30 cmH₂O.
* The sigh pressure was identical in both PEEP steps.

Data CollectionBaseline demographics (age, sex, BMI), comorbidities, and hemodynamics are recorded. At the end of each 15-minute step (baseline and PEEP+3), we perform an end-inspiratory hold and an end-expiratory hold on a tidal assisted breath and measured:

* Plateau pressure (Pplat): Pplat is considered reliable only if the pressure trace is visually stable (flat) during the inspiratory hold.
* Static driving pressure: DP_st = Pplat - PEEP.
* Dynamic driving pressure: DP_dyn = Pressure Support + (ΔP_occ × 0.75), where ΔP_occ is the difference between total PEEP and the low airway pressure during the expiratory-hold maneuver.
* Tidal volume (Vt).
* Respiratory system compliance on tidal assisted breath: Crs_tidal = Vt / DP_st.
* P0.1.
* Occlusion pressure (P_occ).
* Pressure Muscle Index: PMI = P_peak - Pplat.
* Ventilatory Ratio (VR).
* Arterial blood gas (ABG). Compliance During Sigh and S/T IndexCrs during the mandatory sigh (Crs_sigh) is computed at each step using the sigh volume and pressure recorded once the inspiratory flow reaches 0 L/min and airway pressure (Paw) is visually stable.The S/T index is defined as the ratio Crs_sigh / Crs_tidal.Using baseline Crs_tidal, we estimate the sigh-induced volume (mL):V_sigh,expected = (Psigh_peak - PEEP) × Crs_tidal,baseline.We also derive a compliance valid for the pressure range above Pplat up to the sigh pressure ("over-plateau" compliance):Crs_overplat = (Vt_sigh - Vt_tidal) / (Psigh - Pplat).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) receiving PSV with the ventilator's sigh function active.

Exclusion Criteria:

* Clinical contraindication to increasing PEEP
* Hemodynamic instability defined as SOFA cardiovascular score ≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Sigh-to-Assisted Breath Respiratory System Compliance Ratio (Crs_sigh/Crs_assisted) | End of each 15-minute step within a single study session (clinical PEEP; clinical PEEP +3 cmH₂O).
  Ratio of respiratory system compliance at the end of a ventilator-delivered sigh to compliance measured during an inspiratory hold on an assisted tidal breath. This normalized metric indexes recruitability during assisted ventilation; higher values indicate greater recruitability. The primary analysis is the within-patient change in the ratio from clinical PEEP to clinical PEEP +3 cmH₂O.

SECONDARY OUTCOMES:
Patients with unreliable plateau pressure during assisted breaths | Across both 15-minute steps within the single study session.
  Proportion of patients in whom Pplat cannot be reliably measured (non-readable or visually unstable for ≥3 seconds) during inspiratory hold maneuvers in assisted breathing at either study step.
Association between sigh-derived recruitability index and change in respiratory system compliance | End of each 15-minute step within the single study session
  Correlation between the sigh-to-assisted compliance ratio at clinical PEEP and the within-patient change in compliance after PEEP increase

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale Maurizio Bufalini, Cesena, Italy
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Italy

IPD SHARING:
Plan to Share IPD: No
Data may be shared after reasonable request to the Principal investigator.

REFERENCES:
- [Background] Shehabi Y, Chan L, Kadiman S, Alias A, Ismail WN, Tan MA, Khoo TM, Ali SB, Saman MA, Shaltut A, Tan CC, Yong CY, Bailey M; Sedation Practice in Intensive Care Evaluation (SPICE) Study Group investigators. Sedation depth and long-term mortality in mechanically ventilated critically ill adults: a prospective longitudinal multicentre cohort study. Intensive Care Med. 2013 May;39(5):910-8. doi: 10.1007/s00134-013-2830-2. Epub 2013 Jan 24. PMID 23344834
- [Background] Marin-Corral J, Dot I, Boguna M, Cecchini L, Zapatero A, Gracia MP, Pascual-Guardia S, Vila C, Castellvi A, Perez-Teran P, Gea J, Masclans JR. Structural differences in the diaphragm of patients following controlled vs assisted and spontaneous mechanical ventilation. Intensive Care Med. 2019 Apr;45(4):488-500. doi: 10.1007/s00134-019-05566-5. Epub 2019 Feb 21. PMID 30790029
- [Background] Bianchi I, Grassi A, Pham T, Telias I, Teggia Droghi M, Vieira F, Jonkman A, Brochard L, Bellani G. Reliability of plateau pressure during patient-triggered assisted ventilation. Analysis of a multicentre database. J Crit Care. 2022 Apr;68:96-103. doi: 10.1016/j.jcrc.2021.12.002. Epub 2021 Dec 21. PMID 34952477
- [Background] Bastia L, Amendolagine L, Pozzi F, Carenini S, Cipolla C, Curto F, Bellani G, Fumagalli R, Chieregato A. Reliability of Respiratory System Compliance Calculation During Assisted Mechanical Ventilation: A Retrospective Study. Crit Care Med. 2023 Oct 1;51(10):e201-e205. doi: 10.1097/CCM.0000000000005964. Epub 2023 Jun 16. PMID 37326475
- [Background] Mauri T, Grieco DL, Spinelli E, Leali M, Perez J, Chiavieri V, Rosa T, Ferrara P, Scaramuzzo G, Antonelli M, Spadaro S, Grasselli G. Personalized positive end-expiratory pressure in spontaneously breathing patients with acute respiratory distress syndrome by simultaneous electrical impedance tomography and transpulmonary pressure monitoring: a randomized crossover trial. Intensive Care Med. 2024 Dec;50(12):2125-2137. doi: 10.1007/s00134-024-07695-y. Epub 2024 Nov 11. PMID 39527121
- [Background] Jonkman AH, Ranieri VM, Brochard L. Lung recruitment. Intensive Care Med. 2022 Jul;48(7):936-938. doi: 10.1007/s00134-022-06715-z. Epub 2022 May 2. No abstract available. PMID 35499759
- [Background] Moraes L, Santos CL, Santos RS, Cruz FF, Saddy F, Morales MM, Capelozzi VL, Silva PL, de Abreu MG, Garcia CS, Pelosi P, Rocco PR. Effects of sigh during pressure control and pressure support ventilation in pulmonary and extrapulmonary mild acute lung injury. Crit Care. 2014 Aug 12;18(4):474. doi: 10.1186/s13054-014-0474-4. PMID 25113136
- [Background] Patroniti N, Foti G, Cortinovis B, Maggioni E, Bigatello LM, Cereda M, Pesenti A. Sigh improves gas exchange and lung volume in patients with acute respiratory distress syndrome undergoing pressure support ventilation. Anesthesiology. 2002 Apr;96(4):788-94. doi: 10.1097/00000542-200204000-00004. PMID 11964584
- [Background] Albert RK, Jurkovich GJ, Connett J, Helgeson ES, Keniston A, Voelker H, Lindberg S, Proper JL, Bochicchio G, Stein DM, Cain C, Tesoriero R, Brown CVR, Davis J, Napolitano L, Carver T, Cipolle M, Cardenas L, Minei J, Nirula R, Doucet J, Miller PR, Johnson J, Inaba K, Kao L. Sigh Ventilation in Patients With Trauma: The SiVent Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1982-1990. doi: 10.1001/jama.2023.21739. PMID 37877609
- [Background] Mauri T, Eronia N, Abbruzzese C, Marcolin R, Coppadoro A, Spadaro S, Patroniti N, Bellani G, Pesenti A. Effects of Sigh on Regional Lung Strain and Ventilation Heterogeneity in Acute Respiratory Failure Patients Undergoing Assisted Mechanical Ventilation. Crit Care Med. 2015 Sep;43(9):1823-31. doi: 10.1097/CCM.0000000000001083. PMID 25985386